CLINICAL TRIAL: NCT04598334
Title: Investigating the Inflammatory Cytokines and Cytokine Storm Among Bangladeshi Patients With COVID-19: a Prospective, Observational Study
Brief Title: Cytokine Storm Among Bangladeshi Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: PR-20084
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Cytokine Storm, COVID-19
Keywords: Cytokine storm; COVID-19; Bangladesh
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and stool samples will be stored in-80'C following a standard operating procedure for testing stool microbiota and cytokines in blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 positive by RT-PCR: specified number of COVID-19 positive patients will be followed up from admission to outcome (discharge/death/referral). Blood samples will be tested at different time points; cytokines and stool microbiota will be tested at the end of the study and we will analyze the study findings.

SUMMARY:
COVID -19, first reported in Wuhan, China, strikes the world hard as a pandemic by spreading up to 213 countries. Bangladesh is also facing its havoc with the death of 3000 among 229,185 cases at its 141st day. Most are mild cases presenting with influenza-like illness with expected recovery. According to World Health Organization, the overall global case fatality rate is currently estimated to be 2.9%. However, patients having severe or critical illness presenting with severe respiratory distress, ARDS or shock suffer most with mortality rates of 49.0-61.5%. Studies suggest that there are mild or severe cytokine storms in severe patients, which is an important cause of death. An exaggerated and uncontrolled release of pro-inflammatory mediators by an overly activated immune system is known as cytokine storms (CS) or cytokine release syndrome (CRS) which has an important role in the hemodynamic insults seen in very ill COVID-19 patients. This aberrant release of pro-inflammatory cytokines causes lung damage, myocarditis, acute kidney injury, etc. In this study, the investigators aim to estimate the burden of cytokines and their correlation with the magnitude of the severity of COVID-19 illness in Bangladeshi adults.

DETAILED DESCRIPTION:
Background:

1. Burden: COVID -19, first reported in Wuhan, China, strikes the world hard as a pandemic by spreading up to 213 countries. Bangladesh is also facing its havoc with the death of 3000 among 229,185 cases at its 141st day. Most are mild cases presenting with influenza-like illness with expected recovery. According to World Health Organization, the overall global case fatality rate is currently estimated to be 2.9%. However, patients having severe or critical illness presenting with severe respiratory distress, ARDS or shock suffer most with mortality of 49.0-61.5%. Studies suggest that there are mild or severe cytokine storms in severe patients, which is an important cause of death. An exaggerated and uncontrolled release of proinflammatory mediators by an overly activated immune system is termed as cytokine storm (CS). Studies depicting that there might be an important relationship between SARS-CoV-2 and gut microbiota, as a marker to predict ARDS, can corroborate with the disease severity and outcomes of COVID-19.
2. Knowledge gap: Cytokine storm (CS) has an important role in the hemodynamic insults seen in very ill COVID-19 patients. In Bangladesh, no study has been conducted to evaluate the level of cytokines and the gut microbiota in COVID-19 patients presenting with different level of severity and their possible correlation with COVID-19.
3. Relevance: It will explore the role of CS and gut microbiota in COVID-19 illness severity. Thus, the results of the study will improve our knowledge and understanding of the problem, and thereby finding their solutions.

Objectives:

To estimate the burden of 'Cytokine Storm' and its correlation with the magnitude of the severity of COVID-19 illness in Bangladeshi adults.

Methods:

This will be a prospective observational study in adults aged ≥18 years old with COVID-19 having mild /moderate/severe/critical symptoms. The investigators will measure their cytokine (IL 6, TNF-Alpha, and IL1 Beta) levels and investigate gut microbiota in addition to regular laboratory tests at different time points of illness.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years,
2. Informed consent obtained for participation,
3. A mild, moderate or severe (±critical cases) RT-PCR confirmed COVID-19 cases,
4. RT-PCR negative healthy volunteers.

Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The largest diarrheal hospital in the world, the icddr,b Dhaka Hospital admits and treats the general population from Dhaka city with complaints of diarrhea, pneumonia, and malnutrition. For this COVID-19 pandemic, it is also treating its staff and their near relatives in addition to the general patients reporting to the hospital. icddr,b Dhaka hospital manage patients according to clinical condition, and refer patients to appropriate COVID-19 facility if deemed necessary.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
COVID-19 positive participants having high cytokines | Eight months
  The proportion of COVID-19 positive participants having high cytokines during the study period

SECONDARY OUTCOMES:
High cytokine burden and severe COVID-19 | Eight months
  The proportion of participants having both high cytokine burden and severe COVID-19 illness.

OTHER OUTCOMES:
Participants outcome as improved and discharged/referred/deteriorated/death | Six months
  Participants outcome (improved & discharged/referred/deteriorated/death) as percentage
Coagulation profile | Six months
  The proportion of participants having abnormal coagulation profile
Score on chest X-ray | Six months
  The proportion of participants having a poor score on chest X-ray
Gut microbiota | Eight months
  The frequency distribution of different gut microbiota from stool specimen by 16S rRNA sequencing
Three cytokines (IL-6, IL1β, TNF α) in healthy participants | Eight months
  The mean value of cytokines (IL-6, IL1β, TNF α) in healthy participants

CONTACTS AND LOCATIONS:
Overall Officials: Monira Sarmin, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Medicine JHU. COVID-19 Dashboard by the Center for Systems Science and Engineering (CSSE) at Johns Hopkins 2020 [Available from: https://coronavirus.jhu.edu/map.html.
- [Result] IEDCR. COVID-19: Institute of Epidemiology Disease Control and Research; 2020 [Available from: https://www.iedcr.gov.bd/website/index.php/component/content/article/73-ncov-2019.
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Result] National Guidelines on Clinical Management of Coronavirus Disease 2019 (COVID-19). version 7 ed. Government of the People's Republic of Bangladesh: Directorate General of Health Services; 2020.
- [Result] Organization WH. Clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected: interim guidance, 13 March 2020. World Health Organization; 2020.
- [Result] Science Brief: COVID-19 Vaccines and Vaccination. 2021 Sep 15. National Center for Immunization and Respiratory Diseases (NCIRD), Division of Viral Diseases. CDC COVID-19 Science Briefs [Internet]. Atlanta (GA): Centers for Disease Control and Prevention (US); 2020-2023. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK570435/ PMID 34009769
- [Result] Corona virus: Encyclopædia Britannica, Inc./Patrick O'Neill Riley; 2020 [Available from: https://www.britannica.com/science/coronavirus-virus-group.
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Liao D, Zhou F, Luo L, Xu M, Wang H, Xia J, Gao Y, Cai L, Wang Z, Yin P, Wang Y, Tang L, Deng J, Mei H, Hu Y. Haematological characteristics and risk factors in the classification and prognosis evaluation of COVID-19: a retrospective cohort study. Lancet Haematol. 2020 Sep;7(9):e671-e678. doi: 10.1016/S2352-3026(20)30217-9. Epub 2020 Jul 10. PMID 32659214
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- [Result] de Jager W, Bourcier K, Rijkers GT, Prakken BJ, Seyfert-Margolis V. Prerequisites for cytokine measurements in clinical trials with multiplex immunoassays. BMC Immunol. 2009 Sep 28;10:52. doi: 10.1186/1471-2172-10-52. PMID 19785746
- [Result] Teijaro JR, Walsh KB, Rice S, Rosen H, Oldstone MB. Mapping the innate signaling cascade essential for cytokine storm during influenza virus infection. Proc Natl Acad Sci U S A. 2014 Mar 11;111(10):3799-804. doi: 10.1073/pnas.1400593111. Epub 2014 Feb 26. PMID 24572573
- [Result] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Result] Soy M, Keser G, Atagunduz P, Tabak F, Atagunduz I, Kayhan S. Cytokine storm in COVID-19: pathogenesis and overview of anti-inflammatory agents used in treatment. Clin Rheumatol. 2020 Jul;39(7):2085-2094. doi: 10.1007/s10067-020-05190-5. Epub 2020 May 30. PMID 32474885
- [Result] Monteagudo LA, Boothby A, Gertner E. Continuous Intravenous Anakinra Infusion to Calm the Cytokine Storm in Macrophage Activation Syndrome. ACR Open Rheumatol. 2020 May;2(5):276-282. doi: 10.1002/acr2.11135. Epub 2020 Apr 21. PMID 32267081
- [Result] Borthwick LA. The IL-1 cytokine family and its role in inflammation and fibrosis in the lung. Semin Immunopathol. 2016 Jul;38(4):517-34. doi: 10.1007/s00281-016-0559-z. Epub 2016 Mar 21. PMID 27001429
- [Result] Irving K. Acute phase reactants: UpToDate; 2020 [Available from: https://www.uptodate.com/contents/acute-phase-reactants?search=acute%20phase%20reactants&source=search_result&selectedTitle=1~150&usage_type=default&display_rank=1.
- [Result] Sun X, Wang T, Cai D, Hu Z, Chen J, Liao H, Zhi L, Wei H, Zhang Z, Qiu Y, Wang J, Wang A. Cytokine storm intervention in the early stages of COVID-19 pneumonia. Cytokine Growth Factor Rev. 2020 Jun;53:38-42. doi: 10.1016/j.cytogfr.2020.04.002. Epub 2020 Apr 25. PMID 32360420
- [Result] Fu B, Xu X, Wei H. Why tocilizumab could be an effective treatment for severe COVID-19? J Transl Med. 2020 Apr 14;18(1):164. doi: 10.1186/s12967-020-02339-3. PMID 32290839
- [Result] Tanaka T, Narazaki M, Kishimoto T. IL-6 in inflammation, immunity, and disease. Cold Spring Harb Perspect Biol. 2014 Sep 4;6(10):a016295. doi: 10.1101/cshperspect.a016295. PMID 25190079
- [Result] Tobias Herold M, Arnreich C, Hellmuth JC, Matthias Klein M, Tobias Weinberger M. Level of IL-6 predicts respiratory failure in hospitalized symptomatic COVID-19 patients.
- [Result] wikipedia. Tumor necrosis factor 2020 [Available from: https://en.wikipedia.org/wiki/Tumor_necrosis_factor.
- [Result] Gong J, Dong H, Xia QS, Huang ZY, Wang DK, Zhao Y, Liu WH, Tu SH, Zhang MM, Wang Q, Lu FE. Correlation analysis between disease severity and inflammation-related parameters in patients with COVID-19: a retrospective study. BMC Infect Dis. 2020 Dec 21;20(1):963. doi: 10.1186/s12879-020-05681-5. PMID 33349241
- [Result] Wikipedia. Interleukin 1 beta 2020 [Available from: https://en.wikipedia.org/wiki/Interleukin_1_beta.
- [Result] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Result] Kritas SK, Ronconi G, Caraffa A, Gallenga CE, Ross R, Conti P. Mast cells contribute to coronavirus-induced inflammation: new anti-inflammatory strategy. J Biol Regul Homeost Agents. 2020 January-February,;34(1):9-14. doi: 10.23812/20-Editorial-Kritas. PMID 32013309
- [Result] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Result] NIH. COVID-19 treatment guideline, Pharmacologic Interventions [Available from: https://www.covid19treatmentguidelines.nih.gov/critical-care/pharmacologic-interventions/.
- [Result] Tufan A, Avanoglu Guler A, Matucci-Cerinic M. COVID-19, immune system response, hyperinflammation and repurposing antirheumatic drugs. Turk J Med Sci. 2020 Apr 21;50(SI-1):620-632. doi: 10.3906/sag-2004-168. PMID 32299202
- [Result] Hashimoto T, Perlot T, Rehman A, Trichereau J, Ishiguro H, Paolino M, Sigl V, Hanada T, Hanada R, Lipinski S, Wild B, Camargo SM, Singer D, Richter A, Kuba K, Fukamizu A, Schreiber S, Clevers H, Verrey F, Rosenstiel P, Penninger JM. ACE2 links amino acid malnutrition to microbial ecology and intestinal inflammation. Nature. 2012 Jul 25;487(7408):477-81. doi: 10.1038/nature11228. PMID 22837003
- [Result] Turnbaugh PJ, Ley RE, Hamady M, Fraser-Liggett CM, Knight R, Gordon JI. The human microbiome project. Nature. 2007 Oct 18;449(7164):804-10. doi: 10.1038/nature06244. PMID 17943116
- [Result] Lievin-Le Moal V, Servin AL. The front line of enteric host defense against unwelcome intrusion of harmful microorganisms: mucins, antimicrobial peptides, and microbiota. Clin Microbiol Rev. 2006 Apr;19(2):315-37. doi: 10.1128/CMR.19.2.315-337.2006. PMID 16614252
- [Result] Salzman NH, Underwood MA, Bevins CL. Paneth cells, defensins, and the commensal microbiota: a hypothesis on intimate interplay at the intestinal mucosa. Semin Immunol. 2007 Apr;19(2):70-83. doi: 10.1016/j.smim.2007.04.002. Epub 2007 May 7. PMID 17485224
- [Result] Liang J, Sha SM, Wu KC. Role of the intestinal microbiota and fecal transplantation in inflammatory bowel diseases. J Dig Dis. 2014 Dec;15(12):641-6. doi: 10.1111/1751-2980.12211. PMID 25389085
- [Result] Dickson RP, Schultz MJ, van der Poll T, Schouten LR, Falkowski NR, Luth JE, Sjoding MW, Brown CA, Chanderraj R, Huffnagle GB, Bos LDJ; Biomarker Analysis in Septic ICU Patients (BASIC) Consortium. Lung Microbiota Predict Clinical Outcomes in Critically Ill Patients. Am J Respir Crit Care Med. 2020 Mar 1;201(5):555-563. doi: 10.1164/rccm.201907-1487OC. PMID 31973575
- [Result] Meyer NJ, Calfee CS. Novel translational approaches to the search for precision therapies for acute respiratory distress syndrome. Lancet Respir Med. 2017 Jun;5(6):512-523. doi: 10.1016/S2213-2600(17)30187-X. Epub 2017 May 26. PMID 28664850
- [Result] Kyo M, Nishioka K, Nakaya T, Kida Y, Tanabe Y, Ohshimo S, Shime N. Unique patterns of lower respiratory tract microbiota are associated with inflammation and hospital mortality in acute respiratory distress syndrome. Respir Res. 2019 Nov 6;20(1):246. doi: 10.1186/s12931-019-1203-y. PMID 31694652
- [Result] Dickson RP, Singer BH, Newstead MW, Falkowski NR, Erb-Downward JR, Standiford TJ, Huffnagle GB. Enrichment of the lung microbiome with gut bacteria in sepsis and the acute respiratory distress syndrome. Nat Microbiol. 2016 Jul 18;1(10):16113. doi: 10.1038/nmicrobiol.2016.113. PMID 27670109
- [Result] He Y, Wang J, Li F, Shi Y. Main Clinical Features of COVID-19 and Potential Prognostic and Therapeutic Value of the Microbiota in SARS-CoV-2 Infections. Front Microbiol. 2020 Jun 5;11:1302. doi: 10.3389/fmicb.2020.01302. eCollection 2020. PMID 32582134
- [Result] Medicine BSo. COVID-19 management guideline-Bangladesh Model. Dhaka, Bangladesh2020
- [Result] Organization WH. Use of chest imaging in COVID-19 11 June 2020.